CLINICAL TRIAL: NCT05669066
Title: The Effect of Mindful Meditation on Opioid Consumption in Patients Who Undergo Primary Total Hip and Knee Replacement
Brief Title: Meditation and Opioid Consumption in Total Joint Replacement Patients Undergo Primary Total Hip and Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jacob Drew, Assistant Professor of Orthopedic Surgery, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000180
Record Dates: First submitted 2022-06-08; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Arthropathy of Knee; Osteo Arthritis Knee; Osteonecrosis; Meditation; Knee Osteoarthritis; Knee Disease; Knee Injuries; Opioid Use; Opioid Dependence; Opioid Use Disorder
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis, Knee; Knee Injuries; Opioid-Related Disorders | interventions — Mindfulness; Meditation

STUDY DESIGN:
Intervention Model Description: Patients were randomized to 2 groups. The Meditation group or the Control group. The meditation group was asked to meditate 2 times a day, for 2 weeks preoperatively and for 30 days post operatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will undergo a standardized conventional intra-operative and postoperative analgesia regimen. Anesthetic type and postoperative analgesia will be standardized.
- Mindful meditation (Experimental): Start the MM program 2 weeks preoperatively and continue for 30 days post operatively. Study subjects will meet with the meditation instructor for 30 minutes once, 2 weeks prior to surgery, and daily during hospital admission following total joint replacement (TJR). Throughout the intervention period, subjects will be asked to practice daily 15 minutes twice a day, and record their daily meditation experience. Upon discharge from hospital, subjects will receive telephone follow up sessions with the research assistant weekly until 30 days have elapsed. Subjects will be required to show compliance by recording their daily meditation experience in the Daily Meditation Diary (Post-op). At the end of the meditation intervention period, subjects will be asked to provide their feedback in the Patient Satisfaction Survey. Will undergo a standardized, conventional intra-operative postoperative analgesia regimen in addition to the meditation intervention. Anesthetic type will be standardized
  Interventions: Behavioral: Mindful meditation

INTERVENTIONS:
Behavioral: Mindful meditation — Adding mindful meditation to pre- and post-operative care for patients who are having a TKA
  Other Names: meditation; Isha Kriya meditation; Sadhguru meditation
  Arms: Mindful meditation

SUMMARY:
The main purpose of this study is to look at whether meditation techniques can help reduce pain and opioid use after surgery.

DETAILED DESCRIPTION:
Background: The Center for Disease Control identified prescription drug abuse as one of the top 5 current health threats in the US. Orthopedic Surgeons rank among the top 3 prescribers of opioid analgesics. Opioids are commonly used following total knee arthroplasty. Peri- operative protocols have been developed to reduce opioid intake however complications related to opioid analgesics remain problematic resulting in increased morbidity and mortality. There is a pressing need for non-narcotic adjuncts that can minimize /eliminate the use of opioids following elective total knee arthroplasty (TKA). Mind-body techniques including mindful medication (MM) have been demonstrated to reduce pain in acute and chronic disease states.

Purpose: To determine whether mindful meditation, in conjunction with standard analgesic protocols, can impact opioid consumption, pain and function following elective primary TKA.

Methods: a prospective, randomized control trial was conducted in patients aged 18-99 with degenerative joint disease of the knee presenting for primary TKA. Controls received standard perioperative analgesia. In additional to standard analgesia, study patients performed Isha-Krya meditation peri-operatively for 2 weeks followed by 4 weeks post operatively. Outcome measures: opioid consumption, time to discontinue opioids, Pain by Visual Analog Score (VAS), Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) Global Health Short Form, Knee injury and Osteoarthritis Outcome Score (KOOS)

ELIGIBILITY:
Inclusion Criteria:

* • Male and female, ages 18-89 years

  * Narcotic naive patients ("Narcotic naïve" for the purpose of this study will be no history of narcotic tolerance prior to surgery, defined by the FDA as greater than or equal to 60mg oral morphine equivalents per day for 7 days or longer)
  * Scheduled for primary total knee replacement for osteoarthritis
  * Willing to sign informed consent form

Exclusion Criteria:

* • Surgery to be performed for other disease entities (e.g., inflammatory arthritis, post septic arthritis, posttraumatic arthritis or acute fracture)

  * History of narcotic tolerance prior to surgery (defined by the FDA as greater than or equal to 60mg oral morphine equivalents per day for 7 days or longer)
  * Currently taking non-narcotic analgesics other than acetaminophen and non-steroidal anti-inflammatory medications (e.g. Tramadol)
  * History of pain syndromes (e.g., fibromyalgia, complex regional pain syndrome, chronic low back pain)
  * Dementia or other disorder of cognitive function that precludes study consent and/or participation in the MM program
  * In investigator's opinion, unable to complete study tasks over 12-month follow-up period

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 12 months
  visual analog scale (VAS) pain score. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain. A higher score (closer to 10mm) is worse pain and a worse outcome.
Narcotic consumption | 12 months
  Measuring the amount of opioids taken

SECONDARY OUTCOMES:
Length of stay | Recorded at time of discharge (up to 4 days post-operatively)
  Monitoring how long the patient was in the hospital
Discharge to extended care facilities | Recorded at time of discharge (up to 5 days post-operatively)
  Recording where the patient was discharged too
Hospital readmission | 90 days post-operatively
  Recording whether or not the patient was readmitted to the hospital
PROMIS mental health score | 90 days post-operatively
  PROMIS mental health survey. The measures are generic, rather than disease-specific, and use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. It is a survey of 10 questions which gives a physical health and mental health score. The raw global health mental score (4-20) is converted to a mental health T score (16.2-67.7). The higher the score, the better the health outcome.
PROMIS physical health score | 90 days post-operatively
  PROMIS physical health survey. The measures are generic, rather than disease-specific, and use an "In General" item context as it is intended to globally reflect individuals' assessment of their health. It is a survey of 10 questions which gives a physical health and mental health score. The raw global health physical score (4-20) is converted to a physical health T score (16.2-67.7). The higher the score, the better the health outcome.
KOOS Jr Score | 90 days post-operatively
  KOOS JR survey. The KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Drew, MD, Principal Investigator — Beth Israel Deaconess Medical Center 330 Brookline Ave Boston, MA 02215
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Volkow ND, McLellan TA, Cotto JH, Karithanom M, Weiss SR. Characteristics of opioid prescriptions in 2009. JAMA. 2011 Apr 6;305(13):1299-301. doi: 10.1001/jama.2011.401. No abstract available. PMID 21467282
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Nelson AE, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of hip symptoms and radiographic and symptomatic hip osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2009 Apr;36(4):809-15. doi: 10.3899/jrheum.080677. Epub 2009 Mar 13. PMID 19286855
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Young AC, Buvanendran A. Pain management for total hip arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):13-21. doi: 10.3113/jsoa.2014.0013. PMID 24641893
- [Background] Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: a prospective randomized study. J Arthroplasty. 2007 Sep;22(6 Suppl 2):33-8. doi: 10.1016/j.arth.2007.03.034. Epub 2007 Jul 26. PMID 17823012
- [Background] Halawi MJ, Vovos TJ, Green CL, Wellman SS, Attarian DE, Bolognesi MP. Opioid-Based Analgesia: Impact on Total Joint Arthroplasty. J Arthroplasty. 2015 Dec;30(12):2360-3. doi: 10.1016/j.arth.2015.06.046. Epub 2015 Jul 2. PMID 26220104
- [Background] Goesling J, Moser SE, Zaidi B, Hassett AL, Hilliard P, Hallstrom B, Clauw DJ, Brummett CM. Trends and predictors of opioid use after total knee and total hip arthroplasty. Pain. 2016 Jun;157(6):1259-1265. doi: 10.1097/j.pain.0000000000000516. PMID 26871536
- [Background] Simkin DR, Black NB. Meditation and mindfulness in clinical practice. Child Adolesc Psychiatr Clin N Am. 2014 Jul;23(3):487-534. doi: 10.1016/j.chc.2014.03.002. PMID 24975623
- [Background] Rosenzweig S, Greeson JM, Reibel DK, Green JS, Jasser SA, Beasley D. Mindfulness-based stress reduction for chronic pain conditions: variation in treatment outcomes and role of home meditation practice. J Psychosom Res. 2010 Jan;68(1):29-36. doi: 10.1016/j.jpsychores.2009.03.010. PMID 20004298
- [Background] Rangasamy V, Thampi Susheela A, Mueller A, F H Chang T, Sadhasivam S, Subramaniam B. The effect of a one-time 15-minute guided meditation (Isha Kriya) on stress and mood disturbances among operating room professionals: a prospective interventional pilot study. F1000Res. 2019 Mar 26;8:335. doi: 10.12688/f1000research.18446.1. eCollection 2019. PMID 32665843
- [Background] Packiasabapathy S, Susheela AT, Mueller A, Patxot M, Gasangwa DV, O'Gara B, Shaefi S, Marcantonio ER, Yeh GY, Subramaniam B. Guided meditation as an adjunct to enhance postoperative recovery after cardiac surgery: study protocol for a prospective randomized controlled feasibility trial. Trials. 2019 Jan 11;20(1):39. doi: 10.1186/s13063-018-3103-8. PMID 30635064